CLINICAL TRIAL: NCT06914687
Title: Tirellizumab Combined With SOX and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in the Treatment of Peritoneal Metastatic Gastric/Gastroesophageal Junction Adenocarcinoma: A Single-arm, Phase II Clinical Trial (Solids-03)
Brief Title: Efficacy of Tirellizumab Combined With Oral, Intravenous and Abdominal Chemotherapy in Peritoneal Metastatic Gastric/Gastroesophageal Junction Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Fenglin Liu, MD PhD, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOLIDS-03
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Gastric Adenocarcinoma; Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma or Esophageal Carcinoma; Peritoneal Metastasis
Keywords: gastric cancer; Peritoneal Metastasis; Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — tislelizumab; S 1 (combination); Oxaliplatin; Docetaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab plus SOX and HIPEC (Experimental): Tislelizumab, chemotherapy (SOX), and HIPEC(Docetaxel or paclitaxel)
  Interventions: Drug: Tislelizumab; Drug: S-1; Drug: Oxaliplatin; Drug: Docetaxel; Drug: Paclitaxel

INTERVENTIONS:
Drug: Tislelizumab — recombinant humanized anti-PD-1 monoclonal antibody for injection; 200mg ivdrip，d1, q3w
Drug: S-1 — 40~60mg Bid，d1~14, q3w
Drug: Oxaliplatin — 130mg/m2，iv drip for 2h，d1, q3w
Drug: Docetaxel — Docetaxel at a dose of 20 mg/m2 or paclitaxel at a dose of 40 mg/m2 dissolved in 3-5 L of normal saline heated to 43 ± 0.5 °C for HIPEC.(d01-d03,qd,before first cycle of Tislelizumab and SOX)
Drug: Paclitaxel — Paclitaxel at a dose of 40 mg/m2 or docetaxel at a dose of 20 mg/m2 dissolved in 3-5 L of normal saline heated to 43 ± 0.5 °C for HIPEC.(d01-d03,qd,before first cycle of Tislelizumab and SOX)

SUMMARY:
For peritoneal metastatic gastric/gastroesophageal junction adenocarcinoma (cT3-4NanyM1), PD-1 antibody combined with chemotherapy and hyperthermic intraperitoneal chemotherapy (HIPEC) can downstage tumor stage, increase the conversion resection rate, and may improve the long-term survival. Tislelizumab, an anti-PD-1 antibody, has recently been proved in the first- and second-line standard treatment for advanced or metastatic gastric or gastro-oesophageal junction adenocarcinoma.In the subgroup analysis of RATIONALE-305 trial, tislelizumab also showed good efficacy in gastric/gastroesophageal junction adenocarcinoma patients with peritoneal metastasis. Combination of tirellizumab,SOX and HIPEC for peritoneal metastatic gastric/gastroesophageal junction adenocarcinoma could be a novel therapeutic strategy to increase response rate and therapeutic efficacy. This study is a monocenter, single-arm phase 2 clinical trial to evaluate tolerability, safety and efficacy of perioperative tirellizumab in combination with SOX and HIPEC in peritoneal metastatic gastric/gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
The incidence of gastric and gastroesophageal junction adenocarcinoma is increasing, and it is one of the most common malignant tumors in China. Surgery is the only possible way to cure gastric and gastroesophageal junction adenocarcinoma. Peritoneal metastasis is one of the most common modes of spread of gastric cancer. For gastric cancer with peritoneal metastasis, surgical treatment alone can not improve overall survival. Perioperative immunotherapy plus chemotherapy can downstage tumor T and N stage, increase the R0 resection rate, and may improve the long-term survival. Currently, surgical treatment combined with hyperthermic intraperitoneal chemotherapy (HIPEC) and systemic chemotherapy has demonstrated promising outcomes in both the treatment and prevention of peritoneal metastasis in gastric cancer. However, the therapeutic effects of immunotherapy combined with chemotherapy and HIPEC for gastric cancer with peritoneal metastasis remains unclear to date. Combination of perioperative tislelizumab and SOX plus HIPEC for peritoneal metastatic gastric/gastroesophageal junction adenocarcinoma could be a novel therapeutic strategy to increase conversion resection rate and overall survival. This monocenter, single-arm phase 2 clinical trial aims to evaluate the effectiveness of tislelizumab plus SOX and HIPEC regimens in patients with peritoneal metastatic gastric/gastroesophageal junction adenocarcinoma to determine the optimal therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent Patients age 18-75 years Histologically CT/MRI confirmed cT3-4NanyM1 gastric or GEJ adenocarcinoma; Peritoneal metastasis was confirmed by laparoscopy (with or without Krukenberg tumor ) The degree of peritoneal metastasis ≤P1b or PCI≤13 points ECOG 0-1, no surgery contraindications; Expected survival ≥3 months;

Exclusion Criteria:

Prior chemotherapy, radiotherapy, surgery for gastric cancer; Signs of other distant metastases (e.g., liver, lung, bone, supraclavicular lymph, etc.) Significant cardiovascular disease Major surgical procedure within 4 weeks prior to initiation of study treatment Current treatment with anti-viral therapy or HBV Pregnancy or breastfeeding History of malignancy within 5 years prior to screening Present or history of any autoimmune disease or immune deficiency Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) or CTLA-4 agent There are active gastric and duodenal ulcers, ulcerative colitis and other gastrointestinal diseases, or active bleeding in unresectable tumors Poorly controlled hypertension or diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
One year overall survival | From the initiation date of first cycle to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 years

IPD SHARING:
Plan to Share IPD: Undecided